CLINICAL TRIAL: NCT01839357
Title: An Open-label, International, Multicenter, Interventional Study Exploring the Efficacy of Once-daily Oral Rivaroxaban (BAY 59-7939) for the Treatment of Left Atrial/Left Atrial Appendage Thrombus in Subjects With Nonvalvular Atrial Fibrillation or Atrial Flutter
Brief Title: Exploring the Efficacy of Once Daily Oral Rivaroxaban for Treatment of Thrombus in Left Atrial/Left Atrial Appendage in Subjects With Nonvalvular Atrial Fibrillation or Atrial Flutter
Acronym: X-TRA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16320; 2012-001062-15 (EudraCT Number)
Record Dates: First submitted 2013-04-22; First posted 2013-04-24 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2015-12

CONDITIONS: Atrial Fibrillation
Keywords: Rivaroxaban; Oral anticoagulant; Nonvalvular atrial fibrillation; Left atrial thrombus; Transesophageal echocardiography; Thrombus resolution; Stroke; Thromboembolism
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Thromboembolism | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rivaroxaban (Experimental)
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Rivaroxaban 20 mg orally once daily for 6 weeks; subjects with severe to moderate renal impairment (ie, CrCl of 15 to 49 mL/min, inclusive) will receive the adjusted dose of 15 mg orally once daily for 6 weeks in the study.

SUMMARY:
A study for subjects with atrial fibrillation (AF) or atrial flutter who are diagnosed with left atrial (LA) or left atrial appendage (LAA) thrombus. The study will assign subjects to rivaroxaban for treatment of thrombi. The study will measure thrombus outcomes based on echo image and common clinical outcomes such as bleeding and stroke or thromboembolism.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged >/= 18 years
* Hemodynamically stable nonvalvular AF or atrial flutter
* LA/LAA thrombus documented at baseline by transesophageal echocardiography (TEE) up to 72 hours prior to start of study medication
* vitamin K antagonist(s) (VKA)/ new oral anticoagulant(s) (NOAC)-naïve or untreated within 1 month prior to signing of the informed consent form
* VKA pretreated but under ineffective INR levels(<2.0,documented with at least 2 consecutive measurements that are at least 24 hours apart) within last 6 weeks
* Women of childbearing potential and men must agree to use adequate contraception when sexually active

Exclusion Criteria:

* Transient Ischemic Attack within 3 days prior to study inclusion
* Severe, disabling stroke (modified Rankin score of 4-5, inclusive) within 3 months or any stroke within 14 days before the start of study drug
* Acute thromboembolic events or thrombosis (venous/arterial) within the last 14 days prior to study inclusion
* Acute myocardial infarction within the last 14 days prior to study inclusion
* Cardiac-related criteria: Previous intracardiac thrombus, Free-floating ball thrombus, Intracardiac tumor, known left ventricular or aortic thrombus
* Active bleeding or high risk for bleeding contraindicating anticoagulant therapy
* Concomitant drugs/therapies: Indication for anticoagulant therapy for a condition other than nonvalvular AF or atrial flutter (eg, venous thromboembolism). Concomitant use of anticoagulant drugs, including VKA, or factor IIa or factor Xa inhibitors. Chronic aspirin therapy >100 mg or dual antiplatelet therapy. Concomitant use of strong inhibitors of both cytochrome P450 (CYP) 3A4 and P glycoprotein (P-gp), ie, all human immunodeficiency virus protease inhibitors and the following azole antimycotics agents-ketoconazole, itraconazole, voriconazole, and posaconazole-if used systemically
* Concomitant conditions: Childbearing potential without proper contraceptive measures, pregnancy, or breast feeding. Hypersensitivity to investigational treatment. Calculated creatinine clearance (CrCl) < 15 mL/minute at the screening visit. Hepatic disease which is associated with coagulopathy leading to a clinically relevant bleeding risk. Any severe condition that would limit life expectancy to less than 3 months (eg, advanced malignancy, etc.). Planned invasive procedure with potential for uncontrolled bleeding or increased risk of stroke, including major surgery, cardiac catheterization, or cardioversion prior to the end-of-treatment TEE. Inability to take oral medication. Ongoing drug addiction or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-08; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The percentage of subjects with complete resolution of left atrial or left atrial appendage thrombus at the end of treatment | After 6 weeks
  Complete resolution is characterized as the subject is completely thrombus-free confirmed on transesophageal echocardiography

SECONDARY OUTCOMES:
Categories of thrombus outcome in subjects: resolved, reduced, unchanged, enlarged or new | After 6 weeks
The composite number of stroke and non-central nervous system systemic embolism events | Up to 12 weeks
The number of all bleeding events | Up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (25):
- Bulgaria (3):
  - Plovdiv
  - Sofia
  - Varna
- France (4):
  - Créteil
  - Marseille
  - Paris
  - Toulouse
- Germany (4):
  - Hamburg, Hamburg
  - Bonn, North Rhine-Westphalia
  - Leipzig, Saxony
  - Berlin, State of Berlin
- Poland (5):
  - Krakow
  - Lodz
  - Lublin
  - Warsaw
  - Wroclaw
- Russia (3):
  - Moscow
  - Saint Petersburg
  - Saratov
- Turkey (Türkiye) (2):
  - Istanbul
  - Samsun
- Ukraine (4):
  - Donetsk
  - Kiev
  - Odesa
  - Uzhhorod

REFERENCES:
- [Derived] Lip GY, Hammerstingl C, Marin F, Cappato R, Meng IL, Kirsch B, Morandi E, van Eickels M, Cohen A. Rationale and design of a study exploring the efficacy of once-daily oral rivaroxaban (X-TRA) on the outcome of left atrial/left atrial appendage thrombus in nonvalvular atrial fibrillation or atrial flutter and a retrospective observational registry providing baseline data (CLOT-AF). Am Heart J. 2015 Apr;169(4):464-71.e2. doi: 10.1016/j.ahj.2014.12.020. Epub 2015 Jan 6. PMID 25819852